CLINICAL TRIAL: NCT00500617
Title: Identification of Gene Expression Patterns in Circulating Cells That Predict the Presence of Coronary Artery Disease
Brief Title: Personalized Risk Evaluation and Diagnosis (Using Corus CAD or ASGES) in the Coronary Tree
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000004; PREDICT (Other: CardioDx)
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Heart Disease; CAD; CVD; CHD
Keywords: Atherosclerosis; Biological Markers; Molecular Genetics; Gene Expression; GES; CAD; CVD; CHD; Clinical Validity; Precision Medicine; ASGES; CT Angiography; Corus CAD; Coronary angiorgram; Age/Sex/Gene expression Score; Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Disease; Coronary Heart Disease; CTA; PREDICT
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, buffy coat, spun plasma, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- segment 1: Gene discovery blood draw
  Interventions: Diagnostic Test: Corus CAD (ASGES)
- sement 2: Assay development blood draw
  Interventions: Diagnostic Test: Corus CAD (ASGES)
- segment 3: Assay validation blood draw
  Interventions: Diagnostic Test: Corus CAD (ASGES)
- segment 4: Additional assay testing blood draw (Note: post discovery diabetic subjects assigned to this group)
  Interventions: Diagnostic Test: Corus CAD (ASGES)

INTERVENTIONS:
Diagnostic Test: Corus CAD (ASGES) — Age/Sex/Gene Expression Score - ASGES

SUMMARY:
The PREDICT study is to develop and validate a diagnostic blood ASGES (age, sex, gene expression score) or Corus CAD for atherosclerotic coronary artery disease (CAD). The Corus CAD (Age/Sex/Gene Expression score - ASGES) will use quantitative real-time PCR (RT-PCR) to quantify the expression of multiple genes from circulating peripheral blood cells to assess the presence of clinically significant CAD in a patient.

DETAILED DESCRIPTION:
The purpose of the PREDICT study is to develop and validate a diagnostic blood ASGES (age, sex, gene expression score) or Corus CAD for atherosclerotic coronary artery disease (CAD). The Corus CAD (Age/Sex/Gene Expression score - ASGES) will use quantitative real-time PCR (RT-PCR) to quantify the expression of multiple genes from circulating peripheral blood cells to assess the presence of clinically significant CAD in a patient.

This is a prospective, multi-center, observational study. Participation in the study does not alter clinical care. The only procedure required by the protocol is collection of a research blood sample. All other data collected will be in accordance with each participating institution's standard patient care.

The study is divided into four sequential segments with unique subjects and goals: ASGES (Corus CAD) discovery (segment 1), ASGES (Corus CAD) development (segment 2), ASGES (Corus CAD) validation (segment 3), and additional ASGES (Corus CAD) testing (segment 4). The primary analysis will be performed during the third segment of the study using a subset of the enrolled subjects ("primary subjects"). Primary subjects will be defined by additional eligibility criteria beyond the general eligibility criteria required for enrollment in the overall study. The additional, post-enrollment eligibility criteria will be based on clinical and demographic factors that are found during the course of the study to affect the expression of genes used in the ASGES (Corus CAD). Such factors will be identified during gene discovery and algorithm development. The post-enrollment eligibility criteria will be defined prior to the beginning of the ASGES (Corus CAD) validation segment of the study.

In addition, three substudies are planned and will enroll up to 1500 subjects.

* The first substudy will include subjects undergoing cardiac CT angiography (CTA) and aims to determine how gene expression correlates with total coronary atheroma burden, as measured by CTA.
* The second substudy examines sample handling and shipping conditions and does not affect the treatment of the subjects.
* The third substudy will focus on additional algorithm development and validation in a non-diabetic female patient population.

ELIGIBILITY:
Inclusion Criteria:

* Referral for a coronary angiogram (either invasive X-ray angiography or coronary CTA)
* Any one of the following clinical syndromes:

  1. chest pain syndrome, stable angina, or anginal equivalent suggesting myocardial ischemia
  2. low-risk unstable angin, or
  3. asymptomatic individuals with a high probability of CAD

Exclusion Criteria:

* History of myocardial infarction or known CAD
* Current Myocardial Infarct (MI), acute coronary syndrome with high-risk features or unstable angina with high-risk features
* New York Heart Association (NYHA) class III or IV congestive
* Inability to give informed congestive heart failures
* Severe left ventricular systolic dysfunction (LVEF<35%)
* Severe regurgitant or stenotic cardiac valve lesion
* Active or chronic systemic infection
* Rheumatologic, autoimmune or hematologic conditions
* Any organ transplant
* Immunosuppressive therapy
* Chemotherapy in the preceding year
* Major blood or blood product transfusion in the preceding 2 months

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing clinically indicated invasive coronary artery angiogram or CT angiogram.
Sampling Method: Probability Sample
Enrollment: 4350 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Algorithm AUC >0.50 | 30days
  The primary analysis will be performed during the third segment of the study using a subset of the enrolled subjects ("primary subjects"). The primary endpoint for the PREDICT study is a validated algorithm that can accurately classify subjects with and without any coronary artery lesion with a ≥50% diameter stenosis, as measured by Core Laboratory blinded quantitative coronary angiography. In evaluating this endpoint, subjects will be classified as either cases or controls. The endpoint will be assessed by calculating the area under the curve (AUC) for the algorithm score, and testing against an AUC = 0.50 to determine clinical utility, using an alpha level of 0.05 (two-sided).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Monane, MD FACP CMQ, Study Chair — CardioDx
Locations (10):
- United States (10):
  - Alaska Heart Institute, Anchorage, Alaska
  - CV Medical Group Southern California, Beverly Hills, California
  - Scripps HealthCare, La Jolla, California
  - Washington Hospital Medical Center, Washington D.C., District of Columbia
  - Fuqua Heart Center of Atlanta, Atlanta, Georgia
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Allegheny Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain HealthCare, Salt Lake City, Utah

REFERENCES:
- [Result] Rosenberg S, Elashoff MR, Beineke P, Daniels SE, Wingrove JA, Tingley WG, Sager PT, Sehnert AJ, Yau M, Kraus WE, Newby LK, Schwartz RS, Voros S, Ellis SG, Tahirkheli N, Waksman R, McPherson J, Lansky A, Winn ME, Schork NJ, Topol EJ; PREDICT (Personalized Risk Evaluation and Diagnosis in the Coronary Tree) Investigators. Multicenter validation of the diagnostic accuracy of a blood-based gene expression test for assessing obstructive coronary artery disease in nondiabetic patients. Ann Intern Med. 2010 Oct 5;153(7):425-34. doi: 10.7326/0003-4819-153-7-201010050-00005. PMID 20921541
- [Result] Voros S, Elashoff MR, Wingrove JA, Budoff MJ, Thomas GS, Rosenberg S. A peripheral blood gene expression score is associated with atherosclerotic Plaque Burden and Stenosis by cardiovascular CT-angiography: results from the PREDICT and COMPASS studies. Atherosclerosis. 2014 Mar;233(1):284-90. doi: 10.1016/j.atherosclerosis.2013.12.045. Epub 2014 Jan 20. PMID 24529158
- [Result] Beineke P, Fitch K, Tao H, Elashoff MR, Rosenberg S, Kraus WE, Wingrove JA; PREDICT Investigators. A whole blood gene expression-based signature for smoking status. BMC Med Genomics. 2012 Dec 3;5:58. doi: 10.1186/1755-8794-5-58. PMID 23210427
- [Result] Lansky A, Elashoff MR, Ng V, McPherson J, Lazar D, Kraus WE, Voros S, Schwartz RS, Topol EJ. A gender-specific blood-based gene expression score for assessing obstructive coronary artery disease in nondiabetic patients: results of the Personalized Risk Evaluation and Diagnosis in the Coronary Tree (PREDICT) trial. Am Heart J. 2012 Sep;164(3):320-6. doi: 10.1016/j.ahj.2012.05.012. Epub 2012 Jul 24. PMID 22980297
- [Result] Rosenberg S, Elashoff MR, Lieu HD, Brown BO, Kraus WE, Schwartz RS, Voros S, Ellis SG, Waksman R, McPherson JA, Lansky AJ, Topol EJ; PREDICT Investigators. Whole blood gene expression testing for coronary artery disease in nondiabetic patients: major adverse cardiovascular events and interventions in the PREDICT trial. J Cardiovasc Transl Res. 2012 Jun;5(3):366-74. doi: 10.1007/s12265-012-9353-z. Epub 2012 Mar 7. PMID 22396313
- [Result] Elashoff MR, Wingrove JA, Beineke P, Daniels SE, Tingley WG, Rosenberg S, Voros S, Kraus WE, Ginsburg GS, Schwartz RS, Ellis SG, Tahirkheli N, Waksman R, McPherson J, Lansky AJ, Topol EJ. Development of a blood-based gene expression algorithm for assessment of obstructive coronary artery disease in non-diabetic patients. BMC Med Genomics. 2011 Mar 28;4:26. doi: 10.1186/1755-8794-4-26. PMID 21443790
- [Derived] Daniels SE, Beineke P, Rhees B, McPherson JA, Kraus WE, Thomas GS, Rosenberg S. Biological and analytical stability of a peripheral blood gene expression score for obstructive coronary artery disease in the PREDICT and COMPASS studies. J Cardiovasc Transl Res. 2014 Oct;7(7):615-22. doi: 10.1007/s12265-014-9583-3. Epub 2014 Aug 14. PMID 25119856